CLINICAL TRIAL: NCT03280121
Title: Hernia Reduction Prior to Scheduled TIF Completion- The HEURISTIC Study
Brief Title: Hernia Reduction Prior to Scheduled TIF Completion
Acronym: HEURISTIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment and Covid-19
Sponsor: EndoGastric Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D031517
Record Dates: First submitted 2017-09-09; First posted 2017-09-12 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2020-10

CONDITIONS: Fundoplication
Keywords: transoral incisionless

STUDY DESIGN:
Intervention Model Description: Prospective, investigator initiated, multicenter, non-randomized single arm, open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TIF using EsophyX ZR transoral device (Experimental): Transoral incisionless fundoplication which is a minimally invasive treatment for gastroesophageal reflux disease (GERD) using EsophyX ZR transoral device
  Interventions: Device: EsophyX ZR transoral device

INTERVENTIONS:
Device: EsophyX ZR transoral device — TIF

SUMMARY:
Hernia Reduction Prior to Scheduled TIF Completion using EsophyX ZR transoral device

DETAILED DESCRIPTION:
Evaluation of the relative merits, safety and effectiveness of the EsophyX ZR transoral device in performing the standardized TIF 2.0 procedure preceded by laparoscopic Hiatal Hernia repair in PPI-prescribed patients with persistent "troublesome symptoms" per the Montreal consensus definition

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-72 years
2. Dependent upon daily PPIs for > 6 months. Daily use is defined as a double dose, or full dose or half dose taken daily for more than 80% of the total number of days during the proceeding evaluation period
3. Troublesome symptoms, specifically heartburn or regurgitation, while on optimized dose of PPI's Troublesome heartburn or regurgitation symptoms are those which occur a minimum of 2 days a week and are mild to severe in severity
4. Abnormal ambulatory (Bravo) pH study after off PPI therapy for 7 days, i.e. > 5.3% of the time with pH < 4 in a 48-hour monitoring period
5. Normal or near normal esophageal motility (by Upper GI/ esophagram or manometry as required)
6. Pre-enrollment Hiatal Hernia (axial height and transverse dimension) from > 2 cm up to 4 cm inclusive.
7. Patient willing to cooperate with post-operative dietary recommendations and assessment tests at the requisite follow-up visits
8. Signed informed consent Exclusion Criteria

1. BMI > 35 2. Hiatal hernia ≤ 2 and > 4 cm 3. Esophagitis Los Angeles grade C or D 4. Esophageal ulcer 5. Esophageal stricture 6. Long-segment Barretts esophagus (Prague: C > 1, M > 3) 7. Esophageal motility disorder 8. Pregnancy or plans for pregnancy in the next 12 months (in females) 9. Immunosuppression 10. ASA > 2 11. Portal hypertension and/or varices 12. History of previous resective gastric or esophageal surgery, cervical spine fusion, Zenker's diverticulum, esophageal epiphrenic diverticulum, achalasia, scleroderma or dermatomyositis, eosinophilic esophagitis, or cirrhosis 13. Active gastro-duodenal ulcer disease 14. Gastric outlet obstruction or stenosis 15. Severe gastroparesis or delayed gastric emptying confirmed by solid-phase gastric emptying study if patient complains of postprandial satiety during assessment 16. Coagulation disorders 17. Atypical symptoms including gas bloat and dysphagia. 18. Any other presenting condition that in the opinion of the investigator would not make participation in this study in the patient's best interest.

Post Enrollment Exclusion -

1. Inability to repair Hiatal hernia with at least 2cm of intra-abdominal esophagus length.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Murray, MD,FACS, Principal Investigator — Northern Nevada Medical Group
Locations (3):
- United States (3):
  - Elkhart General Hospital, Elkhart, Indiana
  - Aspirus Iron River Hospital, Iron River, Michigan
  - Northern Nevada Medical Center, Sparks, Nevada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were two sites that recruited patients. One was in Iron Mountain. Michigan and one in Sparks, Nevada. The procedures were done in hospitals. The recruitment was from August 18 2018 through February 2019. The study was closed by the sponsor due to slow enrollment.
Groups:
- TIF Using EsophyX ZR Transoral Device: Prospective, investigator initiated, multicenter, non-randomized single arm, open label
Period: Overall Study
Arm/Group | TIF Using EsophyX ZR Transoral Device
Started | 14
Completed | 8
Not Completed | 6
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Not completed — screen failure - 3 hernia too small and 1 pH too low | 4

BASELINE CHARACTERISTICS:
Arm/Group | TIF Using EsophyX ZR Transoral Device
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 62 [36 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: pH Study
Description: Number of Participants with Normalization of Esophageal Acid Exposure. Normalization in esophageal acid exposure is defined by ≤ 5.3% of total time pH < 4 in
Time Frame: 48 hour monitoring period
Measure: Count of Participants; unit: Participants
Groups:
- TIF Using EsophyX ZR Transoral Device-(SINGLE ARM): Transoral incisionless fundoplication which is a minimally invasive treatment for gastroesophageal reflux disease (GERD) using EsophyX ZR transoral device
  EsophyX ZR transoral device: TIF
Arm/Group | TIF Using EsophyX ZR Transoral Device-(SINGLE ARM)
Number analyzed (Participants) | 8
Participants | 6

2. Secondary Outcome: Number of Participants With a Change in Troublesome Symptoms From Baseline
Description: Per Montreal Consensus definition, troublesome symptoms are mild symptoms occurring two (2) or more days per week, or moderate/severe symptoms occurring more than 1 day per week
Time Frame: 6 months
Population: The relatively small number of patients that were willing to come back for follow-up and assessment of outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | TIF Using EsophyX ZR Transoral Device-(SINGLE ARM)
Number analyzed (Participants) | 3
Participants | 3

3. Secondary Outcome: Number of Participants With a Change in PPI Consumption From Baseline to 6 Months
Description: from daily use to occasional use or none at all.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | TIF Using EsophyX ZR Transoral Device-(SINGLE ARM)
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- EsophyX ZR Transoral Device: Transoral incisionless fundoplication which is a minimally invasive treatment for gastroesophageal reflux disease (GERD) using EsophyX ZR transoral device with Hiatal hernias ≤ 2 and > 4 cm.
Arm/Group | EsophyX ZR Transoral Device
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EsophyX ZR Transoral Device (N=14)
Bleeding, hematoma requiring intervention (Gastrointestinal disorders) | 1 (1) — The patient admitted, 10 days post op, for bleeding. Required 2 units of blood. Possibly procedure related but not device related. Husband stated she carried heavy boxes. IRB notified . The issue resolved on 11/17/18.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT03280121/Prot_SAP_ICF_000.pdf